CLINICAL TRIAL: NCT04188236
Title: A Multi-center, Prospective Study to Evaluate the Safety and Performance of a Hernia Blocking System to Prevent Recurrent Lumbar Disc Herniation
Brief Title: Safety and Performance of a Hernia Blocking System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-RA1-2018-01
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Disk Herniated Lumbar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hernia Blocking System — Hernia Blocking System device implanted during a lumbar discectomy procedure

SUMMARY:
Prospective, multi-center, single-arm clinical study to assess the performance of an Hernia Blocking System in preventing clinically symptomatic recurrent lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 75 years of age.
* Posterolateral disc herniation at one level between L4 and S1 with radiographic confirmation (CT and/or MRI) of neural compression.
* At least six weeks of failed conservative treatment prior to surgery, including physical therapy, use of anti-inflammatory medications at maximum specified dosage and/or administration of epidural/facet injections.
* Minimum posterior disc height of 5 mm at the index level.
* Radiculopathy with positive straight leg raise test.
* ODI score of at least 40/100.
* Subjects who are able to give voluntary informed consent to participate in the clinical investigation and from whom consent has been obtained.
* Subject is able and willing to comply with the protocol requirements.

Exclusion Criteria:

* Spondylolisthesis and/or instability at the index level.
* Foraminal, extra-foraminal or central disc herniation.
* Subject has clinically compromised vertebral bodies in the lumbosacral region due to any traumatic, neoplastic, metabolic, or infectious pathology.
* Subject has scoliosis of greater than 20 degrees (both angular and rotational).
* Less than 20 mm of interpedicular distance in the spinal canal at the index level.
* Grossly distorted anatomy due to congenital abnormalities.
* Deformation that affect the posterior corners of the vertebra at the index level (e.g., osteophytes).
* Endplate irregularities that, in the judgment of the surgeon, could affect the device implantation.
* Prior surgery at the index lumbar vertebral level.
* Radiological confirmation of severe facet joint disease or degeneration.
* Patients diagnosed or at a high risk of osteoporosis (such as postmenopausal women and patients receiving long-term treatment with corticosteroids) who present a bone densitometry DXA T-score of less than -2.0 at the index level.
* Cauda equina syndrome.
* Fever, leucocytosis and/or systemic or localized active infection.
* Systemic inflammation and/or inflammation at the implantation site.
* Any metabolic bone disease.
* Insulin-dependent diabetes mellitus.
* Peripheral neuropathy.
* Active hepatitis, AIDS or HIV.
* Rheumatoid arthritis or other autoimmune disease.
* Active or history of any invasive malignancy; patients with curatively-treated malignancies who have been disease-free for at least 5 years are eligible.
* Active tuberculosis or history of tuberculosis in the past 3 years.
* Immunologically suppressed patients.
* Current anticoagulation therapy, unless anticoagulation therapy can be suspended for surgery.
* Patients who have received medication (e.g., methotrexate, alendronate) that interferes with bone mineral metabolism within 4 weeks of the planned date of the index surgery.
* Suspected or known allergies or intolerance to the implant materials.
* Any condition that precludes the use of general anesthesia.
* Any condition that precludes the surgical procedure.
* Any contraindication for MRI or CT scan.
* Class III obesity: Body mass index ≥ 40.
* Current alcohol or recreational drug dependency.
* Pregnant or interested in becoming pregnant in the following 24 months.
* Breastfeeding.
* Life expectancy less than 2 years.
* Subject is currently participating or has participated in the previous 4 weeks in any other interventional clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically symptomatic recurrent lumbar disc herniation | 24 months

SECONDARY OUTCOMES:
The incidence and type of all adverse events (AE) and serious adverse events (SAE). | 6 weeks, 6 months, 12 months, and 24 months
Incidence of clinically asymptomatic recurrent disc herniation | 6 months, 12 months, and 24 months
Disc height maintenance [mm] related to baseline | 6 weeks, 6 months, 12 months, and 24 months
Change in leg and low back pain assessed by NRS (numeric rating scale), related to baseline | 6 weeks, 6 months, 12 months, and 24 months
  0-10 NRS
Change in Low back related disability according to the Oswestry Disability Index (ODI), related to baseline | 6 weeks, 6 months, 12 months, and 24 months
The change in quality of life according to EQ-5D-5L, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
The change in the patient work status, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
The change in patient neurological status: straight leg raise test, reflexes, motor muscle strength and sensory neurological evaluations, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
The change in the kinematics of the intervertebral disc at the index level, compared to baseline | 6 weeks, 6 months, 12 months, and 24 months
The change in the disc degeneration (Pfirrmann scale), compared to baseline | 6 months, 12 months, and 24 months
The change in the endplate lesions (MODIC scale), compared to baseline | 6 months, 12 months, and 24 months

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital QuirónSalud Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catala I, Roldan H, Fernandez-Carballal C, Dominguez-Alonso C, Alvarez-Galovich L, Godino O. A new hernia blocking system prevents lumbar disc herniation recurrence and disc degeneration: 2 years results of a multicentric clinical investigation. Brain Spine. 2025 Dec 3;6:105898. doi: 10.1016/j.bas.2025.105898. eCollection 2026. PMID 41492501
- [Derived] Godino O, Fernandez-Carballal C, Catala I, Moreno A, Rimbau JM, Alvarez-Galovich L, Roldan H. A new hernia blocking system to prevent recurrent lumbar disc herniation: surgical technique, intraoperative findings and six-months post-operative outcomes. Eur Spine J. 2025 Mar;34(3):1123-1133. doi: 10.1007/s00586-024-08595-x. Epub 2024 Dec 8. PMID 39648196